CLINICAL TRIAL: NCT03368300
Title: Epidemiology and Pathophysiology of Parkinsonism in the Caribbeans
Acronym: CAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBM-PAP-2011/86
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Atypical Parkinsonism
Keywords: progressive supranuclear palsy; Caribbean atypical Parkinsonism; Annona Muricata
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Intervention Model Description: The primary aim of this study is to estimate the frequency and to characterize clinically atypical parkinsonism in the French West Indies and Guyana.
  This study has been designed as epidemiological, multicentric transversal descriptive and longitudinal prospective study with biological collection and post-mortem neuropathological sub-study of brain tissue.
Masking Description: Not masking, 2 groups parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Parkinson's patient
  Interventions: Other: Clinical and biological exam
- witnesses: without parkinson's disease (Other): Subjects without parkinson's disease
  Interventions: Other: Clinical and biological exam

INTERVENTIONS:
Other: Clinical and biological exam — The study will include a clinical, neuropsychological, oculomotor, food intake and environmental exposure assessment. Blood samples will be taken to constitute a library of plasma, DNA and serum. The harvesting of samples will be part of a subsequent study. Consent for possible post-mortem neuropathological analysis will be proposed.
  All the patients accepting it will be followed by a 5-year longitudinal follow-up. The longitudinal follow-up bi-annual and then annual will include a clinical evaluation, a questionnaire of dependence and a questionnaire of monitoring of exposure to certain environmental factors
  All controls must answer a questionnaire of environmental exposure factors, oculomotor test, and blood sample (3 collections: DNA, serum, plasma).

SUMMARY:
The primary aim of this study is to estimate the frequency and to characterize clinically atypical parkinsonism in the French West Indies and Guyana.

DETAILED DESCRIPTION:
An atypical akineto-rigid parkinsonian syndrome, unresponsive to L-dopa has been evidenced in Guadeloupe. Abnormally frequent, this progressive supranuclear palsy (PSP)-like syndrome represents a new clinical entity. Unlike in classical PSP 70% of patients have myoclonus, 59% hallucinations, 78% REM sleep behavior disorders. Oculomotor pattern differs from classical PSP suggesting that cortical dysfunction predominates over brainstem impairments. Neuropathological examination in four patients has shown a widespread accumulation of the tau protein in the basal ganglia, the midbrain and cortical areas.

This syndrome has been associated to the regular consumption of food products derived from plants of the Annonaceae family, more specifically Annona Muricata (soursop), suggesting a toxic origin. We have already confirmed the neurotoxic potential of the lipophilic mitochondrial complex I inhibitor annonacin, the major acetogenin in Annona muricata. This class of compounds is specific to Annonaceae. Nanomolar concentrations of annonacin induce the death of dopaminergic neurons in culture, by impairment of energy production. Chronic systemic intoxication of rats with annonacin causes neuronal damage in the same brain regions that are damaged in patients with atypical parkinsonism. These results greatly suggest that the consumption of annonacea might contribute to the pathogenesis of the disease. The H1 subhaplotype in tau gene associated with PSP in Caucasians did not confer risk for PSP-like atypical parkinsonism in Guadeloupe.

ELIGIBILITY:
Inclusion Criteria:

* Pour les patients :

  1. Patient ou tiers responsable ayant reçu une information sur l'étude et ayant signé le consentement éclairé
  2. Patient âgé de plus de 18 ans
  3. Patient consultant en neurologie ou en gériatrie pour symptomatologie parkinsonienne ou pour troubles cognitifs évocateurs d'une démence à corps de Lewy
  4. Patient domicilié aux Antilles-Guyane

     Pour les témoins :
  5. Conjoint ou accompagnant ayant reçu une information sur l'étude et ayant signé le consentement éclairé
  6. Personne âgée de plus de 18 ans
  7. Personne ne présentant pas de pathologie d'allure neurodégénérative (Parkinson, démence notamment)
  8. Personne domiciliée aux Antilles-Guyane

Exclusion Criteria:

Pour les patients :

1. Syndrome parkinsonien secondaire (post-traumatique, vasculaire, iatrogène, post encéphalitique)
2. Patient non affilié au régime de sécurité sociale
3. En cas de difficulté de suivi le patient sera exclu de l'étude longitudinale

Pour les témoins :

1. Personnes présentant des troubles cognitifs ou un syndrome parkinsonien diagnostiqué.
2. Patient non affilié au régime de sécurité sociale -

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2012-08-03 (Actual); Primary Completion 2018-08-03 (Estimated); Study Completion 2023-08-03 (Estimated)

PRIMARY OUTCOMES:
to estimate the frequency and to characterize clinically atypical parkinsonism in the French West Indies and Guyana | At the end of the Period of inclusion, around 5-6 years
  Collection of :
  administrative and socioeconomic data, medical consultation with video recording , recording oculomotor to the atypical

SECONDARY OUTCOMES:
to compare the proportion of atypical forms within parkinsonian syndromes; | At the end of the Period of inclusion, around 5-6 years
  Collection of :
  administrative and socioeconomic data, medical consultation with video recording , recording oculomotor to the atypical neuropsychological balance assessment ,
  1. Clinical diagnostic criteria
  2. Compilation of functional indicators of motor and cognitive autonomy and Collection of intercurrent medical events
  3. Food and exposure questionnaire
  4. Neuropsychological assessment
  5. Recording of oculomotor movements and Post-mortem analysis
  6. biological collection (plasma, DNA, serum)
to characterize the entity "Parkinson-dementia complex" described in Guadeloupe ; to characterize the entity "Parkinson-dementia complex" described in Guadeloupe ; | Through study completion, an average of 11 years
  Compilation of functional indicators of motor and cognitive autonomy and Collection of intercurrent medical events.
  Collection of :
  administrative and socioeconomic data, medical consultation with video recording , recording oculomotor to the atypical neuropsychological balance assessment ,
to determine the natural history of typical and atypical forms of parkinsonism by following a cohort of the incident cases only; | Through study completion, an average of 11 years
  Neuropsychological assessment Food and exposure survey
to determine the implication of a toxic alimentary factor in the etiopathogenesis of atypical forms and compare the results in the 3 areas (Guadeloupe, Guyane, Martinique); | Through study completion, an average of 11 years
  Neuropsychological assessment Food and exposure survey
to determine the latency of cognitive decline in idiopathic Parkinson's disease in the 3 areas ; | Through study completion, an average of 11 years, post-mortem analysis after death if applicable
  Recording of oculomotor movements and Post-mortem analysis (sampling of blood and cutaneous biopsy to establish a collection of biological samples)
to constitute a biological collection (plasma, DNA, serum). | At the end of the Period of inclusion, around 5-6 years
  biological collection (plasma, DNA, serum)

CONTACTS AND LOCATIONS:
Overall Officials: Annie LANNUZEL, PU-PH, Study Director — University Hospital of Guadeloupe; Régine EDRAGAS, PH, Principal Investigator — University Hospital of Martinique; Dominique MARNET, PH, Principal Investigator — : University Hospital of Guyana
Locations (2):
- University Hospital of Guyana, Cayenne, French Guiana
- University Hospital of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No